CLINICAL TRIAL: NCT06569329
Title: Bacterial Reduction After Supplementary Disinfection Procedures in Infected Root Canals
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abhishek Parolia (Other)
Responsible Party: Sponsor-Investigator, Abhishek Parolia, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 202402221
Record Dates: First submitted 2024-08-19; First posted 2024-08-26 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-08

CONDITIONS: Dental Pulp Necroses
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- GentleWave System Root Canal Therapy (Experimental): Sterile paper points will be inserted into the root canal at 3 time points: (i) before instrumentation, (ii) after washing the canal with 10% sodium thiosulfate, and (iii) after the GentleWave System root canal therapy has been completed. The paper points will collect bacteria, which will be analyzed via real-time Polymerase Chain Reaction to assess bacterial counts.
  Interventions: Device: GentleWave System Root Canal Therapy
- EdgePro Laser Root Canal Therapy (Experimental): Sterile paper points will be inserted into the root canal at 3 time points: (i) before instrumentation, (ii) after washing the canal with 10% sodium thiosulfate, and (iii) after the EdgePro Laser root canal therapy has been completed. The paper points will collect bacteria, which will be analyzed via real-time Polymerase Chain Reaction to assess bacterial counts.
  Interventions: Device: EdgePro Laser Root Canal Therapy
- The ProUltra Piezo Ultrasonic with EndoUltra Tips Root Canal Therapy (Experimental): Sterile paper points will be inserted into the root canal at 3 time points: (i) before instrumentation, (ii) after washing the canal with 10% sodium thiosulfate, and (iii) after the ProUltra Piezo Ultrasonic with EndoUltra Tips root canal therapy has been completed. The paper points will collect bacteria, which will be analyzed via real-time Polymerase Chain Reaction to assess bacterial counts.
  Interventions: Device: The ProUltra Piezo Ultrasonic with EndoUltra Tips Root Canal Therapy

INTERVENTIONS:
Device: GentleWave System Root Canal Therapy — This device has 510k market approval for its intended use within this study.
  Arms: GentleWave System Root Canal Therapy
Device: EdgePro Laser Root Canal Therapy — This device has 510k market approval for its intended use within this study.
  Arms: EdgePro Laser Root Canal Therapy
Device: The ProUltra Piezo Ultrasonic with EndoUltra Tips Root Canal Therapy — This device has 510k market approval for its intended use within this study.
  Arms: The ProUltra Piezo Ultrasonic with EndoUltra Tips Root Canal Therapy

SUMMARY:
The purpose of this study is to understand the effect that 3 different types of root canal procedures have on bacteria.

DETAILED DESCRIPTION:
Sample Size Calculation Sample size was calculated by STATISTICA v8.0 software (StatSoft, Tulsa, OK, USA), that demonstrated 23 teeth per group are needed to show a 5% difference in bacterial levels at 90% power. Considering possible losses, ninety adult subjects will be selected.

Case Selection and Eligibility Criteria Participants will be recruited at the Endodontic Clinic at the University of Iowa. The inclusion criteria will be patients 18 years or older, teeth with intact pulp chamber walls, no response to cold and electric pulp testing and apical periodontitis.

Teeth with vital pulp, incomplete root formation, extensive crown destruction, previous endodontic treatment or intervention (pulp debridement), acute/ chronic apical abscess, internal or external resorption, non-odontogenic facial pain, periodontal probing deeper than 4 mm, advanced untreated periodontal disease or recent periodontal surgery, teeth with mobility score > 2, fracture or visible crack, patients with diabetes or immune-compromised conditions, patients who received systemic antibiotics within the last three months, or taking corticosteroids, and pregnancy will be excluded.

Study Intervention Root canal samples will be taken under strict asepsis, as described by Rodrigues et al. (21). Operative field will be disinfected using 3% hydrogen peroxide and 3% NaOCl under rubber dam isolation. Once the access cavity is prepared, 10% sodium thiosulfate solution will be injected into the pulp chamber, and the sterility control (SC) will be taken from the access cavity walls' internal surfaces using sterile paper points. This sample will be transferred aseptically to a cryotube containing RNA later (Ambion, Austin, TX) and stored at -20°C.

The first sample (S1) will be taken as the baseline quantity of bacteria before chemomechanical preparation. One ml of 10% sodium thiosulfate solution will be injected into the canal, and a sterile paper point will be introduced up to that length for 1 minute, transferred in cryotubes containing RNA later, and stored at -20°C.

The root canal will be shaped and cleaned using rotary endodontic instruments up to size 35/.04, with periodic irrigation with 5 mL of 3% NaOCl between each instrumentation. After apical preparation, the canal will be dried with sterile paper points and then washed with 1 mL of 10% sodium thiosulfate for 1 minute to inactivate NaOCl. After that, a second sample (S2) will be collected and stored as described for S1.

Teeth specimens will be randomly assigned to three groups (n=30) according to the type of supplementary disinfection approaches used: (1) GWS, (2) LAI, and (3) UAI. These devices will be used as stated above in phase 1 of this study. After using supplementary disinfection approaches, a third sample (S3) will be collected from the root canal and stored as described above for S1 and S2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of pulp necrosis with apical periodontitis (AP) confirmed by pulp tests, clinical and radiographic evidence.
* Tooth with no response to cold and electric pulp testing (done at screening).
* Single canalled premolars with intact pulp chamber walls.
* Patient must be 18 years of age or older

Exclusion Criteria:

* Teeth with vital pulp.
* Teeth with incomplete root formation (immature with apical periodontitis).
* Teeth with extensive crown destruction.
* Teeth with previous endodontic treatment or intervention (pulp debridement).
* Teeth with acute/ chronic apical abscess.
* Teeth with internal or external resorption.
* Teeth with non-odontogenic facial pain.
* Teeth with periodontal pockets deeper than 4 mm.
* Teeth with advanced untreated periodontal disease or recent periodontal surgery.
* Teeth with mobility score greater than 2.
* Teeth with a fracture or visible crack.
* Patients with diabetes or immune compromised conditions.
* Patients who received systemic antibiotics within the last 3 months.
* Patients taking corticosteroids.
* Patients who are pregnant.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of the changes in the bacterial count at various time points during the root canal procedure. | Baseline (pre-intervention) and during the intervention and immediately after the intervention
  Sterile paper points will be inserted into the root canal in order to collect bacteria. Real-time Polymerase Chain Reaction will be used to assess the bacterial counts.

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Parolia, PhD, MDS, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa College of Dentistry and Dental Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No